CLINICAL TRIAL: NCT07235215
Title: Effects of Vivatlac Synbiotic in Patients With Irritable Bowel Syndrome - A Randomized, Double-blind, Placebo-Controlled, 36 Weeks Clinical Trial
Brief Title: Vivatlac in Irritable Bowel Syndrome II (ViIBS2)
Acronym: ViIBS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kalisz 2025-01 ViIBS Trial II
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; Vivatlac synbiotic; ViIBS2 trial; synbiotic
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized allocation of verum or placebo group of similar size
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Capsule containing maize starch with identical appearance as verum. One capsule taken per day before bedtime. Treatment duration 36 weeks.
  Interventions: Dietary Supplement: Placebo
- Vivatlac Synbiotic (Experimental): Vivatlac Synbiotic for 36 weeks. One capsule containing a mixture of nine different probiotic bacteria with a total amount of 4.5 x 10^9 colony forming units and 63 mg of fructooligosaccharides. One capsule taken per day before bedtime. Treatment duration 36 weeks.
  Interventions: Dietary Supplement: Vivatlac Synbiotic

INTERVENTIONS:
Dietary Supplement: Vivatlac Synbiotic — Vivatlac Synbiotic containing a total of 4.5 x 10^9 colony forming units (CFU) of nine different probiotic bacteria. Probiotic bacteria strains and their CFU amount per capsule are: Lactococcus lactis Ll-23, 9.00 x 10^8 CFU; Lactobacillus helveticus SP 27, 9.00 x 10^8 CFU; Bifidobacterium longum Bl-05, 6.75 x 10^8 CFU; Bifidobacterium longum ES1, 4.50 x 10^8 CFU; Lacticaseibacillus rhamnosus Lr-32, 4.50 x 10^8 CFU; Streptococcus thermophiles St-21, 4.50 x 10^8 CFU; Lacticaseibacillus casei Lc-11, 2.25 x 10^8 CFU; Lactiplantibacillus plantarum Lp-115, 2.25 x 10^8 CFU; Bifidobacterium bifidum Bb-02, 2.25 x 10^8 CFU. As a prebiotic component each capsule contains 63 mg of fructooligosaccharides.
  Arms: Vivatlac Synbiotic
Dietary Supplement: Placebo — Capsule containing maize starch with identical appearance as verum.
  Arms: Placebo

SUMMARY:
Multi-center,randomized, double-blind, placebo-controlled, 36 weeks trial investigating the effects of a nine-strain synbiotic (Vivatlac Synbiotikum) in IBS patients

DETAILED DESCRIPTION:
The study design is a multi-centre, randomized, double-blind, placebo controlled clinical trial in patients diagnosed with IBS. Diagnosis of IBS with the World Gastroenterology Organisation's IBS questionnaire for health care providers. Assessment of severity of IBS by using the IBS Severity of Symptoms Scale (IBS-SSS). IBS patients with moderate to severe IBS will be included into the study (IBS-SSS ≥ 175). A four weeks screening phase is used to evaluate patients' IBS symptoms and stool characteristics using a patient diary.

The screening phase is followed by treatment with one capsule per day of a nine-strain synbiotic (Vivatlac® Synbiotikum) or with an identical looking placebo for thirty-six weeks.

Each capsule of Vivatlac® Synbiotikum contains a total of 4.5 x 10^9 colony forming units (CFU) of nine different probiotic bacteria. Probiotic bacteria strains and their CFU amount per capsule are: Lactococcus lactis Ll-23, 9.00 x 10^8 CFU; Lactobacillus helveticus SP 27, 9.00 x 10^8 CFU; Bifidobacterium longum Bl-05, 6.75 x 10^8 CFU; Bifidobacterium longum ES-1, 4.50 x 10^8 CFU; Lacticaseibacillus rhamnosus Lr-32, 4.50 x 10^8 CFU; Streptococcus thermophiles St-21, 4.50 x 10^8 CFU; Lacticaseibacillus casei Lc-11, 2.25 x 10^8 CFU; Lactiplantibacillus plantarum Lp-115, 2.25 x 10^8 CFU; Bifidobacterium bifidum Bb-02, 2.25 x 10^8 CFU. In addition, each capsule contains 68 mg of fructooligosaccharides (FOS).

Treatment effects will be assessed by using the IBS-Severity Scoring System (IBS-SSS), before the start of treatment and after 4, 8, 12, 24, and 36 weeks of treatment. Changes of IBS severity will be assessed by using the IBS-Global Improvement Scale (IBS-GIS), before the start of treatment and after 4, 8, 12, 24, and 36 weeks of treatment. Patients will be assessed for IBS relief by using the IBS-Adequate Relief scale (IBS-AR), before the start of treatment and after 4, 8, 12, 24, and 36 weeks of treatment. Stool form characteristics will be assessed with the Bristol Stool Form Scale, before the start of treatment and after 4, 8, 12, 24, and 36 weeks treatment. Quality of life (QoL) will be assessed before the start of treatment and after 12 and 36 weeks of treatment using the IBS-QoL questionnaire. Emotional suppression will be assessed before the start of treatment and after 12 and 36 weeks of treatment using the Courtauld Emotional Control Scale (CECS).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed for Irritable Bowel Syndrome using the IBS questionnaire for Health Care Providers of the World Global Gastroenterology Organization
* IBS-SSS ≥ 175 points

Exclusion Criteria:

* patients currently taking products containing probiotics or have taken this kind of products during the last 3 months
* patients currently taking antibiotics or have taken antibiotics during the last 3 months
* patients having a concurrent severe illness (malignancies, uncontrolled hypertension or diabetes, hepatic, renal or cardiac dysfunctions, serious neurological disorders, psychosis, respiratory disorders such as asthma or COPD, hyper- or hypothyroidism
* patients having chronic bowel disorders other than IBS, including inflammatory bowel disease, gastroenteritis, stomach and duodenal cancer, celiac disease
* patient being pregnant, lactating, or planning to become pregnant during the next 9 months
* patient being diagnosed to have a lactose intolerance
* patients using motility drugs or dietary fiber supplements withing 2 weeks before study start
* patient taking anti-coagulant medication
* patients have participated in another clinical trial within the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Severity of IBS using the IBS-Severity Scoring System (IBS-SSS) | Measured at enrollment into treatment phase, and after 12, and 36 weeks of treatment.
  IBS-Severity Scoring System is a 5-question survey that asks: 1. the severity of abdominal pain, 2. frequency of abdominal pain, 3. severity of abdominal distention, 4.dissatisfaction with bowel habit, and 5. interference with quality of life over the past 10 days. Subjects respond to each question on a 100-point visual analogue scale. Each of the five question generates a maximum score of 100 point, and total scores can range from 0-500 with higher scores indicating severe symptoms. A decrease of 50 points is associated with a clinically meaningful improvement.
Changes of IBS severity using the IBS Global Improvement Scale (IBS-GIS) | Measured after 12, and 36 weeks of treatment.
  Patients answer the question "Have you felt any change in the severity of your symptoms over the past 7 days compared to how you felt before the medicine was given?
  The answers are recorded based on the 7-point scale:
  * I feel that the symptoms have worsened significantly
  * I feel that the symptoms have moderately worsened
  * I feel that the symptoms have slightly worsened
  * I feel no change
  * I feel a slight improvement
  * I feel moderate improvement
  * I feel significant improvement IBS-GIS score indicates: improvement if is >4 or worsening if is<4, no change if is 4
Changes in adequate relief of IBS-symptoms (IBS-AR) | Measured after 12, and 36 weeks of treatment.
  IBS-Adequate Relief (IBS-AR) is a dichotomous single item that asks participants "Over the past week (7 days) have you had adequate relief of your IBS symptoms? The answer is YES or NO.

SECONDARY OUTCOMES:
Changes of stool form characteristics (Bristol Stool Form Scale) | Measured at enrollment into treatment phase, and after 4, 8, 12, 24 , and 36 weeks of treatment.
  Type of stools assessed using the Bristol Stool Scale. Bristol Scale is designed to classify faeces into seven groups: type 1-2 indicate constipation, type 3-4 are "normal" stools; type 5-7 indicate diarrhea.
IBS-Quality of Life Measure (IBS-QOL) | Measured at enrollment into treatment phase, and after 12, and 36 weeks of treatment.
  The IBS-QOL is a patient self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. The IBS-QOL consists of 34 items. Each of the items can be responded by selecting from a five-point (1-5) Likert response scale.
  The scoring procedure comprises 2 steps. In the first step a raw total score is determined by summing the individual answers (1-5). Thereafter the raw sum is transformed into a 0-100 scale.
  The formula for the transformation is:
  Score = (Sum of items) - (lowest possible raw score) / Possible raw score range × 100. "Sum of items" = sum of scores to all 34 items of the scale, "Lowest possible raw score" = if someone answers the minimum (e.g. 1) to all items, "Possible raw score range" = (maximum raw score - minimum raw score).
  A higher final score (closer to 100) indicates a poorer QOL related to IBS, lower scores a better QOL.
Changes of Emotional Suppression (Courtauld Emotional Control Scale, CECS) | Measured at enrollment into treatment phase, and after 12, and 36 weeks of treatment.
  The CECS comprises 21 statements divided into three subscales. Each subscale contains seven statements that concern the manner of showing depression, anxiety, and anger. By marking the most suitable answer, respondents assess how oftern they express emotions in a way provided in the questionnaire on a four-point scale from "almost never" - one point to "almost always" four points. The sum of the results in each subscale can range from 7-28 points. A general emotional control coefficient is calculated by adding the scores of the three subscales. The general emotional control coefficient can range from 21 to 84 points. The higher the score, the more supressed emotions are.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Piatek, Prof. Dr., Principal Investigator — The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz
Locations (3):
- Poland (3):
  - District Hospital Jarocin, Jarocin
  - GP Clinic Spitalna, Jarocin
  - GP Clinic Wroclawska, Jarocin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piatek J, Krauss H, Ciechelska-Rybarczyk A, Bernatek M, Wojtyla-Buciora P, Sommermeyer H. In-Vitro Growth Inhibition of Bacterial Pathogens by Probiotics and a Synbiotic: Product Composition Matters. Int J Environ Res Public Health. 2020 May 11;17(9):3332. doi: 10.3390/ijerph17093332. PMID 32403297
- [Background] Sommermeyer H, Pituch HM, Wultanska D, Wojtyla-Buciora P, Piatek J, Bernatek M. Inhibition of Quinolone- and Multi-Drug-Resistant Clostridioides Difficile Strains by Multi Strain Synbiotics-An Option for Diarrhea Management in Nursing Facilities. Int J Environ Res Public Health. 2021 May 30;18(11):5871. doi: 10.3390/ijerph18115871. PMID 34070727
- [Background] Piatek J, Sommermeyer H, Bernatek M, Ciechelska-Rybarczyk A, Oleskow B, Mikkelsen LS, Barken KB. Persistent infection by Salmonella enterica servovar Typhimurium: are synbiotics a therapeutic option? - a case report. Benef Microbes. 2019 Mar 13;10(2):211-217. doi: 10.3920/BM2018.0080. Epub 2018 Dec 21. PMID 30574800
- [Background] Sommermeyer H, Piatek J. Synbiotics as Treatment for Irritable Bowel Syndrome: A Review. Microorganisms. 2024 Jul 21;12(7):1493. doi: 10.3390/microorganisms12071493. PMID 39065261
- [Background] Sommermeyer H, Chmielowiec K, Bernatek M, Olszewski P, Kopczynski J, Piatek J. Results from a Cross-Sectional Observational Study Examining Irritable Bowel Syndrome Patients Six Months After Finishing Their Participation in the ViIBS Trial. Nutrients. 2024 Nov 15;16(22):3911. doi: 10.3390/nu16223911. PMID 39599697
- [Background] Sommermeyer H, Chmielowiec K, Bernatek M, Olszewski P, Kopczynski J, Piatek J. Effectiveness of a Balanced Nine-Strain Synbiotic in Primary-Care Irritable Bowel Syndrome Patients-A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2024 May 16;16(10):1503. doi: 10.3390/nu16101503. PMID 38794741